CLINICAL TRIAL: NCT07075822
Title: Effect of Tapioca-based FiberSMART® Compared to a Glucose Challenge or Water Control on Postprandial Glycemia in Healthy Subjects: An Acute Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INQUIS Clinical Research (Industry)
Collaborators: Anderson Advanced Ingredients (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: INQ-2522
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Demonstrate That the Postprandial Glucose Response of FiberSMART is Consistent With the Response Expected From a Dietary Fiber
Keywords: dietary fiber, postprandial glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FiberSMART® (Experimental): 20g of FiberSMART® dissolved in 250ml of water
  Interventions: Other: 20g of FiberSMART®
- Dextrose (Active Comparator): 20g of dextrose dissolved in 250g of water
  Interventions: Other: 20g of Dextose
- Water Control (Placebo Comparator): 250g of water
  Interventions: Other: Water Control

INTERVENTIONS:
Other: 20g of FiberSMART® — 20g of FiberSMART® dissolved in 250g of water
  Arms: FiberSMART®
Other: 20g of Dextose — 20g of dextrose dissolved in 250g of water
  Arms: Dextrose
Other: Water Control — 250g of water
  Arms: Water Control

SUMMARY:
The goal of this clinical trial is to learn whether a novel tapioca-based soluble fiber, FiberSMART®, affects blood glucose levels after consumption in healthy adult volunteers.

The main questions it aims to answer are:

Does FiberSMART® raise postprandial (after-meal) blood glucose levels? Is the blood glucose response to FiberSMART® different from that of dextrose or water?

Researchers will compare participants' blood glucose responses after consuming 20g of FiberSMART® to their responses after consuming 20g of dextrose or a water control to see if FiberSMART® results in a lower postprandial glucose rise than the dextrose challenge and is no different from the water challenge. Demonstrating the FiberSMART acts like a dietary fiber.

Participants will:

Visit the clinic on three separate mornings after an overnight fast Consume either 20g of FiberSMART® or 20g of dextrose or a water control Undergo 8 finger-prick blood tests over 2 hours to measure blood glucose levels

ELIGIBILITY:
Inclusion Criteria:

* Subjects are healthy adult males and non-pregnant females. Subjects must be eligible to receive income in Canada. Family members of staff and/or staff that have no responsibilities/tasks on this particular trial may be subjects

Exclusion Criteria:

* age less than 18 years;
* any known food allergies or intolerances to the investigational product;
* medications known to affect glucose tolerance -but stable doses of oral contraceptives, acetylsalicylic acid, thyroxin, vitamins and mineral supplements or drugs to treat hypertension or osteoporosis are acceptable;
* known history of diabetes mellitus or the use of anti-hyperglycemic drugs or insulin to treat diabetes and related conditions;
* any major medical or surgical events requiring hospitalization within the preceding 3 months;
* the presence of disease or drug(s) which influence digestion and absorption of nutrients;
* the short-term use of systemic steroids or atypical antipsychotics (<4 weeks) (all of which have major effects on glucose and metabolism and body fat distribution)
* any other medications or conditions which might, in the opinion of the Medical Director of INQUIS Clinical Research Ltd. (INQUIS), either 1) make participation dangerous to the subject or to others, or 2) affect the results;
* any subject who cannot or will not comply with the experimental procedures or do not follow INQUIS safety guidelines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Blood Glucose iAUC | 2 hours post-prandial
  Determine the 2 hour iAUC of FiberSMART® and compare it to the iAUC of dextrose (positive control) and water (negative control). Incremental area under the blood glucose curve (iAUC) will be calculated using the trapezoid rule, ignoring the area beneath the baseline.

SECONDARY OUTCOMES:
Posprandial glucose levels at each time point | 2 hour postprandial
  Compare the blood glucose levels at each time point after consuming 20g FiberSMART® or 20g of dextrose (positive control) or water (negative control).
Glucose Peak Height | 2 hours post-prandial
  Determine the blood glucose peak height (mmol/L) after consuming 20g FiberSMART® and compare it to the blood glucose peak height after consuming 20g of dextrose (positive control) or water (negative control).
Glucose Tmax | 2 hour postprandial
  Determine the time to maximum postprandial glucose level glucose peak height (mmol/L) after consuming 20g FiberSMART® and compare it to the blood glucose peak height after consuming 20g of dextrose (positive control) or water (negative control).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Wolever, MD, PhD, Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No